CLINICAL TRIAL: NCT03821103
Title: Incentivizing Buprenorphine-Naloxone Initiation in Emergency Departments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: American College of Medical Toxicology (Other); Blue Cross Blue Shield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 832359
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Opioid Use

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard training arm (Experimental): The standard training arm will consist of (1) in-person training with pre- and post-session knowledge and attitude assessment, (2) three month post-session knowledge and attitude assessment and (3) self-report of first-time buprenorphine-naloxone Emergency Department administration within 3 month study period.
  Interventions: Behavioral: Training
- Behavioral economic enhanced arm (Experimental): The behavioral economic enhanced training arm will consist of (1) in-person training with pre- and post-session knowledge and attitude assessment, (2) three month post-session knowledge and attitude assessment and (3) self-report of first-time buprenorphine-naloxone Emergency Department administration within 3 month study period in addition to an opt-out invitation, loss-framed incentivization, and weekly tailored text message-based reminders
  Interventions: Behavioral: Training; Behavioral: Behavioral economic enhanced arm

INTERVENTIONS:
Behavioral: Training — The training includes of (1) in-person training with pre- and post-session knowledge and attitude assessment, (2) three month post-session knowledge and attitude assessment and (3) self-report of first-time buprenorphine-naloxone Emergency Department (ED) administration within 3 month study period
Behavioral: Behavioral economic enhanced arm — Behavioral economic enhancement includes an opt-out invitation, loss-framed incentivization, weekly tailored text based reminders
  Arms: Behavioral economic enhanced arm

SUMMARY:
This study seeks to test standard and behavioral economic-enhanced training strategies to bolster first-time Emergency Department-initiated buprenorphine-naloxone administration among Emergency Department providers.

DETAILED DESCRIPTION:
Philadelphia is experiencing a significant opioid crisis. Through this novel pilot study, critical training about opioid use disorder and medication-assisted treatment with buprenorphine-naloxone will be provided to emergency providers and changes in clinical practice will be incentivized in order to optimize treatment engagement for patients with opioid use disorder in the Emergency Department.

Participants will be invited to participate in a brief in-person training session, will receive a pre- and post-session knowledge and attitude assessment, and will be invited to self-report first-time buprenorphine-naloxone Emergency Department administration within the 3 month study period.

Participants will be randomized to one of two arms: standard training arm and behavioral economic enhanced arm. The standard training arm will receive the aforementioned intervention. The behavioral economic enhanced arm will additionally receive an opt-out invitation, loss-framed incentivization, and weekly tailored text message-based reminders.

Endpoints of interest include retained knowledge and change in provider attitudes regarding Emergency department buprenorphine-naloxone administration and treatment following training and again at 3 months, and first-time Emergency department administration of buprenorphine-naloxone.

ELIGIBILITY:
Inclusion Criteria:

* Residents and Advanced Practice Providers and attending clinicians working in emergency departments in Pennsylvania.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Change in Emergency Department initiated buprenorphine-naloxone treatment | One year
  Measuring number of providers who have initiated at least one first dose of buprenorphine-naloxone

SECONDARY OUTCOMES:
Training Attendance | First week
  Measure the number of clinicians who attend the training with the incentive.
Change in attitude about buprenorphine-naloxone Questionaire | Three months
  The scale is not a validated tool. It is a construct to measure attitudes about buprenorphine-naloxone.
  It is a Likert scale 1-5, 1 being strongly disagree and 5 being strongly agree. Higher values signify more favorable outcomes.

OTHER OUTCOMES:
Retained knowledge of buprenorphine-naloxone treatment Questionaire | Three months
  Compare retention of knowledge and assessment from before and after the training in the two arms.The scale is not a validated tool. It is a construct of questions to measure retained knowledge about buprenorphine-naloxone initiation.
  The scale is a percentage of questions answered correctly. Minimum score is 0% and maximum score is 100%.
  Higher values signify more favorable outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanmarie Perrone, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khatri UG, Lee K, Lin T, D'Orazio JL, Patel MS, Shofer FS, Perrone J. A Brief Educational Intervention to Increase ED Initiation of Buprenorphine for Opioid Use Disorder (OUD). J Med Toxicol. 2022 Jul;18(3):205-213. doi: 10.1007/s13181-022-00890-7. Epub 2022 Apr 12. PMID 35415804